CLINICAL TRIAL: NCT06171711
Title: Exposure Therapy for Anorexia Nervosa Pilot Trial
Brief Title: Exposure Therapy Study In Adults With Eating Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Jamal Essayli, Assistant Professor of Pediatrics and Psychiatry & Behavioral Health, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23573
Record Dates: First submitted 2023-12-05; First posted 2023-12-15 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Eating Disorders; Anorexia Nervosa
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa | interventions — Implosive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exposure Therapy (Experimental): Exp-AN will effectively target anxiety related to eating and weight gain via inhibitory learning, and improve treatment outcomes.
  Interventions: Behavioral: Exposure Therapy

INTERVENTIONS:
Behavioral: Exposure Therapy — The proposed study will explore whether Exp-AN works via inhibitory learning (i.e., decreasing anxious beliefs and increasing anxiety tolerance) and/or between-session habituation (i.e., decreasing anxiety levels across therapy sessions), and the importance of targeting anxiety about eating versus weight gain. Results will provide information about the degree to which all three mechanisms of action (i.e., changes in anxiety ratings, anxious beliefs, and tolerance of anxiety) predict improved AN symptomatology across both treatments. Research that discovers whether specific treatments (e.g., Exp-AN) work in the way the investigators think they do (e.g., by increasing tolerance of anxiety), and whether modifying intervention targets (e.g., tolerance of anxiety) helps people get better (e.g., reduced AN symptomatology), will ultimately lead to more personalized, mechanism-based, and effective treatments (Insel 2014; Insel et al., 2010).

SUMMARY:
The current proposal will evaluate the feasibility, acceptability, and preliminary efficacy of Exposure Therapy for anorexia nervosa (AN) spectrum disorders (Exp-AN), an innovative treatment rooted in principles of inhibitory learning. Exp-AN will target anxiety about both eating and weight gain by combining in vivo (i.e., in real life) and imaginal (i.e., mental) exposure in novel ways (e.g., eating a feared food while listening to a recording describing fears about weight gain).

DETAILED DESCRIPTION:
The current proposal will evaluate the feasibility, acceptability, and preliminary efficacy of Exposure Therapy for anorexia nervosa (AN) Spectrum Disorders (Exp-AN), an innovative treatment rooted in principles of inhibitory learning. Exp-AN will target anxiety about both eating and weight gain by combining in vivo (i.e., in real life) and imaginal (i.e., mental) exposure in novel ways (e.g., eating a feared food while listening to a recording describing fears about weight gain).

The central hypothesis is that Exp-AN will effectively target anxiety related to eating and weight gain via inhibitory learning, and improve treatment outcomes. The investigator will test two aims:

Aim 1. Evaluate the feasibility, acceptability, and preliminary efficacy of Exp-AN.

Hypothesis 1.1: Exp-AN will be feasible, with satisfactory levels of recruitment (≥50%) and retention (≥75%).

Hypothesis 1.2: Participants will engage in Exp-AN, as measured by completion of the five treatment modules (≥80%) and therapy homework (≥60%).

Hypothesis 1.3: Participants will rate all five Exp-AN modules as acceptable.

Hypothesis 1.4: Exp-AN will result in increases in BMI and decreases in AN symptomatology.

Aim 2. Investigate Exp-AN's mechanisms of action, and if mechanisms are associated with positive outcomes.

Hypothesis 2.1: Exp-AN will result in decreases in anxiety between sessions, decreases in anxious beliefs, and increases in anxiety tolerance.

Hypothesis 2.2: Changes in anxiety ratings, anxious beliefs, and tolerance of anxiety will be associated with weight gain and reduced AN symptomatology.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be English speakers, ages 17 - 65 years, of all genders, with AN-spectrum disorders, defined as a diagnosis of AN, atypical AN, or AN in partial remission.

   1. Participants with AN, atypical AN, and AN in partial remission share the same DSM-5 criteria, with the exception of criterion A: "Significantly low body weight."
   2. Individuals with atypical AN are weight suppressed, but not "objectively" underweight (e.g., someone who experiences rapid weight loss from a BMI of 27 to 21). Those with AN in partial remission are partially or fully weight restored (e.g., after stepping down from an inpatient setting), but continue to experience significant AN behaviors (e.g., food avoidance) and/or cognitions (e.g., fear of weight gain).
   3. Diagnoses will be determined using the Structured Clinical Interview for DSM-5 - Research Version (SCID-5-RV).93 All participants in this study will be monitored by a Penn State Health medical provider.
2. All individuals who are deemed to be, or become, unsafe by their supervising medical provider will be admitted to our hospital or another facility for medical stabilization.

Exclusion Criteria:

1. Participants will be excluded if they are below 18 years of age.
2. Those identified as non-English speakers will be excluded due to lack of funding to translate the measures to other languages.
3. Individuals with other EDs (e.g., bulimia nervosa) will be excluded.
4. Participants will be excluded if they are:

   a.at high risk for suicide i.Suicide risk will be determined using the Columbia Suicide Severity Rating Scale (CSSRS) screen. The CSSRS will be administered by the study coordinator when they initially meet with the participant for Session 0 (see section 7 of this protocol), and at the start of every weekly session with the study therapist. The study coordinator and study therapists will be trained by the PI to adhere to a Suicide Assessment Protocol. This protocol will state that all participants who report high suicide risk should be sent by an ambulance to our institution's emergency department.

   b.pregnant determined by verbal verification (the study coordinator will ask participants if they are pregnant when completing the eligibility checklist and/or during the informed consent process).

   c. Meet DSM-5 criteria for a psychotic disorder and/or have an intellectual disability.

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Structured Clinical Interview for DSM-5-Research Version (SCID-5-RV) | Admission-Baseline (Week 0)
  The Structured Clinical Interview for DSM-5-Research Version (SCID-5-RV) is comprehensive, including most disorders, subtypes severity, and course specifiers. The instrument provides a diagnostic process to covers the DSM-5 diagnoses most commonly seen in clinical setting such as depressive and bipolar disorders; schizophrenia spectrum and other psychotic disorders; substance use disorders; anxiety disorders (panic disorder, agoraphobia, social anxiety disorder, generalized anxiety disorder); obsessive-compulsive disorder; posttraumatic stress disorder; attention-deficit/hyperactivity disorder, eating disorders and adjustment disorder. It also screens for 17 additional DSM-5 disorders.
Demographic Form | Admission-Baseline (Week 0)
  The Demographic Form is a 10-item self-report questionnaire. It was designed to assess information about the participant's age, race/ethnicity, past medical history, and eating disorder history.
Food Phobia Survey | Admission-Baseline (Week 0)
  The Food Phobia Survey is a 360-item self-report questionnaire. It was designed to assess participant's frequency, fear, guilt, appeal to food, and behaviors associated with a diagnosis of an eating disorder. The scores of items are calculated and range from 0 to 5. The higher rating indicates a higher frequency, fear, guilt, and appeal to food.
Eating Disorder Examination - Self-Report Questionnaire (EDE-Q) | Admission-Baseline (Week 0)
  The Eating Disorder Examination Questionnaire (EDE-Q) is a 28-item self-report questionnaire. It was designed to assess the range, frequency, and severity of behaviors associated with a diagnosis of an eating disorder. A total score is obtained by summing the four subscales scores and dividing the total by the number of subscales. The score of items are calculated and range from 0 to 36. The higher score indicate greater ED symptoms.
Fear of Food Measure (FOFM) | Admission-Baseline (Week 0)
  The Fear of Food Measure (FORM) is a 23-item self-report questionnaire. It examines the participant's severity of behaviors associated with a diagnosis of an eating disorder. Each item is scored on a 1-7 scale. The questionnaire range from 23 to 161 meaning 23: no fear of food and 161 meaning severe fear of food.
Body Shape Questionnaire (BSQ) | Admission-Baseline (Week 0)
  The BSQ is a self-reported measurement of the body shape concerns typical of bulimia nervosa and anorexia nervosa. The questionnaire has 34 items scored from 0 to 6 points (least and most impaired, respectively), with the sum of the questions giving a range from 0 to 204. The higher score indicates greater concerns about body shape.
Clinical Impairment Assessment (CIA) | Admission-Baseline (Week 0)
  The Clinical Impairment Assessment Questionnaire (CIA) is a 16-item self-report measure of the severity of psychosocial impairment due to eating disorder features and focuses on the past 28 days. The 16 items cover impairment in domains of life that are typically affected by eating disorder psychopathology: mood and self-perception, cognitive functioning, interpersonal functioning, and work performance. The responses are scored 0,1,2 and 3, with a higher rating indicating a higher level of impairment. The total range is between 0 and 48.
Eating Disorder Fear Questionnaire (EDFQ) | Admission-Baseline (Week 0)
  The Eating Disorder Fear Questionnaire (EDFQ) is a 20-item self-report questionnaire. It examines the participant's severity of behaviors associated with a diagnosis of an eating disorder. The response range between 1 to 7 with a total range of 20 to 140. The higher rating indicates a higher severe impairment.
Treatment Acceptability Questionnaire | Admission-Baseline (Week 0)
  The Treatment Acceptability Questionnaire is a 10-item self-report questionnaire. It examines the participants' perspective on the modules in the exposure therapy. The response range between 1 to 7, with a total range of 10 to 70. The higher rating indicates a higher rating of treatment acceptability.
Eating Disorder Examination - Self-Report Questionnaire (EDE-Q) | Session 5 (Week 5)
  The Eating Disorder Examination Questionnaire (EDE-Q) is a 28-item self-report questionnaire. It was designed to assess the range, frequency, and severity of behaviors associated with a diagnosis of an eating disorder. A total score is obtained by summing the four subscales scores and dividing the total by the number of subscales. The score of items are calculated and range from 0 to 36. The higher score indicate greater ED symptoms.
Fear of Food Measure (FOFM) | Session 5 (Week 5)
  The Fear of Food Measure (FORM) is a 23-item self-report questionnaire. It examines the participant's severity of behaviors associated with a diagnosis of an eating disorder. Each item is scored on a 1-7 scale. The questionnaire range from 23 to 161 meaning 23: no fear of food and 161 meaning severe fear of food.
Body Shape Questionnaire (BSQ) | Session 5 (Week 5)
  The BSQ is a self-reported measurement of the body shape concerns typical of bulimia nervosa and anorexia nervosa. The questionnaire has 34 items scored from 0 to 6 points (least and most impaired, respectively), with the sum of the questions giving a range from 0 to 204.The higher score indicates greater concerns about body shape.
Clinical Impairment Assessment (CIA) | Session 5 (Week 5)
  The Clinical Impairment Assessment Questionnaire (CIA) is a 16-item self-report measure of the severity of psychosocial impairment due to eating disorder features and focuses on the past 28 days. The 16 items cover impairment in domains of life that are typically affected by eating disorder psychopathology: mood and self-perception, cognitive functioning, interpersonal functioning, and work performance. The responses are scored 0,1,2 and 3, with a higher rating indicating a higher level of impairment. The total range is between 0 and 48.
Eating Disorder Fear Questionnaire (EDFQ) | Session 5 (Week 5)
  The Eating Disorder Fear Questionnaire (EDFQ) is a 20-item self-report questionnaire. It examines the participant's severity of behaviors associated with a diagnosis of an eating disorder. The response range between 1 to 7 with a total range of 20 to 140. The higher rating indicates a higher severe impairment.
Treatment Acceptability Questionnaire | Session 5 (Week 5)
  The Treatment Acceptability Questionnaire is a 10-item self-report questionnaire. It examines the participants' perspective on the modules in the exposure therapy. The response range between 1 to 7, with a total range of 10 to 70. The higher rating indicates a higher rating of treatment acceptability.
Eating Disorder Examination - Self-Report Questionnaire (EDE-Q) | Session 10 (Week 10)
  The Eating Disorder Examination Questionnaire (EDE-Q) is a 28-item self-report questionnaire. It was designed to assess the range, frequency, and severity of behaviors associated with a diagnosis of an eating disorder. A total score is obtained by summing the four subscales scores and dividing the total by the number of subscales. The score of items are calculated and range from 0 to 36. The higher score indicate greater ED symptoms.
Fear of Food Measure (FOFM) | Session 10 (Week 10)
  The Fear of Food Measure (FORM) is a 23-item self-report questionnaire. It examines the participant's severity of behaviors associated with a diagnosis of an eating disorder. Each item is scored on a 1-7 scale. The questionnaire range from 23 to 161 meaning 23: no fear of food and 161 meaning severe fear of food.
Body Shape Questionnaire (BSQ) | Session 10 (Week 10)
  The BSQ is a self-reported measurement of the body shape concerns typical of bulimia nervosa and anorexia nervosa. The questionnaire has 34 items scored from 0 to 6 points (least and most impaired, respectively), with the sum of the questions giving a range from 0 to 204.The higher score indicates greater concerns about body shape.
Clinical Impairment Assessment (CIA) | Session 10 (Week 10)
  The Clinical Impairment Assessment Questionnaire (CIA) is a 16-item self-report measure of the severity of psychosocial impairment due to eating disorder features and focuses on the past 28 days. The 16 items cover impairment in domains of life that are typically affected by eating disorder psychopathology: mood and self-perception, cognitive functioning, interpersonal functioning, and work performance. The responses are scored 0,1,2 and 3, with a higher rating indicating a higher level of impairment. The total range is between 0 and 48.
Eating Disorder Fear Questionnaire (EDFQ) | Session 10 (Week 10)
  The Eating Disorder Fear Questionnaire (EDFQ) is a 20-item self-report questionnaire. It examines the participant's severity of behaviors associated with a diagnosis of an eating disorder. The response range between 1 to 7 with a total range of 20 to 140. The higher rating indicates a higher severe impairment.
Treatment Acceptability Questionnaire | Session 10 (Week 10)
  The Treatment Acceptability Questionnaire is a 10-item self-report questionnaire. It examines the participants' perspective on the modules in the exposure therapy. The response range between 1 to 7, with a total range of 10 to 70. The higher rating indicates a higher rating of treatment acceptability.
Eating Disorder Examination - Self-Report Questionnaire (EDE-Q) | Session 15 (Week 15)
  The Eating Disorder Examination Questionnaire (EDE-Q) is a 28-item self-report questionnaire. It was designed to assess the range, frequency, and severity of behaviors associated with a diagnosis of an eating disorder. A total score is obtained by summing the four subscales scores and dividing the total by the number of subscales. The score of items are calculated and range from 0 to 36. The higher score indicate greater ED symptoms.
Fear of Food Measure (FOFM) | Session 15 (Week 15)
  The Fear of Food Measure (FORM) is a 23-item self-report questionnaire. It examines the participant's severity of behaviors associated with a diagnosis of an eating disorder. Each item is scored on a 1-7 scale. The questionnaire range from 23 to 161 meaning 23: no fear of food and 161 meaning severe fear of food.
Body Shape Questionnaire (BSQ) | Session 15 (Week 15)
  The BSQ is a self-reported measurement of the body shape concerns typical of bulimia nervosa and anorexia nervosa. The questionnaire has 34 items scored from 0 to 6 points (least and most impaired, respectively), with the sum of the questions giving a range from 0 to 204.The higher score indicates greater concerns about body shape.
Clinical Impairment Assessment (CIA) | Session 15 (Week 15)
  The Clinical Impairment Assessment Questionnaire (CIA) is a 16-item self-report measure of the severity of psychosocial impairment due to eating disorder features and focuses on the past 28 days. The 16 items cover impairment in domains of life that are typically affected by eating disorder psychopathology: mood and self-perception, cognitive functioning, interpersonal functioning, and work performance. The responses are scored 0,1,2 and 3, with a higher rating indicating a higher level of impairment. The total range is between 0 and 48.
Eating Disorder Fear Questionnaire (EDFQ) | Session 15 (Week 15)
  The Eating Disorder Fear Questionnaire (EDFQ) is a 20-item self-report questionnaire. It examines the participant's severity of behaviors associated with a diagnosis of an eating disorder. The response range between 1 to 7 with a total range of 20 to 140. The higher rating indicates a higher severe impairment.
Treatment Acceptability Questionnaire | Session 15 (Week 15)
  The Treatment Acceptability Questionnaire is a 10-item self-report questionnaire. It examines the participants' perspective on the modules in the exposure therapy. The response range between 1 to 7, with a total range of 10 to 70. The higher rating indicates a higher rating of treatment acceptability.
Eating Disorder Examination - Self-Report Questionnaire (EDE-Q) | Discharge_Session 20 (Week 20)
  The Eating Disorder Examination Questionnaire (EDE-Q) is a 28-item self-report questionnaire. It was designed to assess the range, frequency, and severity of behaviors associated with a diagnosis of an eating disorder. A total score is obtained by summing the four subscales scores and dividing the total by the number of subscales. The score of items are calculated and range from 0 to 36. The higher score indicate greater ED symptoms.
Fear of Food Measure (FOFM) | Discharge_Session 20 (Week 20)
  The Fear of Food Measure (FORM) is a 23-item self-report questionnaire. It examines the participant's severity of behaviors associated with a diagnosis of an eating disorder. Each item is scored on a 1-7 scale. The questionnaire range from 23 to 161 meaning 23: no fear of food and 161 meaning severe fear of food.
Body Shape Questionnaire (BSQ) | Discharge_Session 20 (Week 20)
  The BSQ is a self-reported measurement of the body shape concerns typical of bulimia nervosa and anorexia nervosa. The questionnaire has 34 items scored from 0 to 6 points (least and most impaired, respectively), with the sum of the questions giving a range from 0 to 204.The higher score indicates greater concerns about body shape .
Clinical Impairment Assessment (CIA) | Discharge_Session 20 (Week 20)
  The Clinical Impairment Assessment Questionnaire (CIA) is a 16-item self-report measure of the severity of psychosocial impairment due to eating disorder features and focuses on the past 28 days. The 16 items cover impairment in domains of life that are typically affected by eating disorder psychopathology: mood and self-perception, cognitive functioning, interpersonal functioning, and work performance. The responses are scored 0,1,2 and 3, with a higher rating indicating a higher level of impairment. The total range is between 0 and 48.
Eating Disorder Fear Questionnaire (EDFQ) | Discharge_Session 20 (Week 20)
  The Eating Disorder Fear Questionnaire (EDFQ) is a 20-item self-report questionnaire. It examines the participant's severity of behaviors associated with a diagnosis of an eating disorder. The response range between 1 to 7 with a total range of 20 to 140. The higher rating indicates a higher severe impairment.
Treatment Acceptability Questionnaire | Discharge_Session 20 (Week 20)
  he Treatment Acceptability Questionnaire is a 10-item self-report questionnaire. It examines the participants' perspective on the modules in the exposure therapy. The response range between 1 to 7, with a total range of 10 to 70. The higher rating indicates a higher rating of treatment acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Jamal Essayli, Principal Investigator — Penn State University
Locations (1):
- 905 W Govener Rd, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No